CLINICAL TRIAL: NCT00022022
Title: Docetaxel In Second-Line Treatment Of Advanced Non-Small-Cell Lung Cancer - The Distal Study
Brief Title: Docetaxel in Treating Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale per lo Studio e la Cura dei Tumori (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068702; ITA-INTN-DISTAL; EU-20103
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which chemotherapy regimen is more effective in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare two different docetaxel regimens in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the quality of life of patients with stage IIIB or IV non-small cell lung cancer treated with 2 different schedules of docetaxel as second-line therapy.
* Compare the toxicity of these regimens in these patients.
* Compare the response rate, time to progression, and survival of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, ECOG performance status (0 vs 1 vs 2), response to prior chemotherapy (partial or complete response vs stable disease vs progressive disease), and prior cisplatin-containing chemotherapy regimen (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV on day 1. Treatment continues every 3 weeks for a maximum of 6 courses.
* Arm II: Patients receive docetaxel IV weekly for 6 weeks. Treatment continues every 8 weeks for a maximum of 2 courses.

Quality of life is assessed at baseline and days 22 and 43-56 for arm I, and at baseline and days 22 and 43 for arm II.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer (NSCLC)

  * Metastatic supraclavicular lymphadenopathy or malignant pleural effusion
  * Progressive disease
  * Must have received prior chemotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN) AST and ALT no greater than 1.25 times ULN

Renal:

* Creatinine no greater than 1.25 times ULN

Cardiovascular:

* No prior or concurrent cardiovascular disease that would preclude study

Pulmonary:

* See Disease Characteristics
* No prior or concurrent pulmonary disease that would preclude study

Other:

* No prior or other concurrent illness or medical condition that would preclude study
* No other prior malignancy except adequately treated carcinoma in situ of the cervix or nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior docetaxel
* At least 3 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed
* No concurrent radiotherapy

Surgery:

* Prior radical surgery for NSCLC allowed
* Concurrent palliative surgery allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2000-12

PRIMARY OUTCOMES:
Quality of life
Toxicity
Response rate
Time to progression
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, MD, Study Chair — Istituto Nazionale per lo Studio e la Cura dei Tumori
Locations (16):
- Italy (16):
  - Istituto Di Ricovero E Cura A Carattere Scientifico, Bari
  - Azienda Ospedaliena G. Rummo, Benevento
  - Ospedale Cardarelli - Campobasso, Campobasso
  - Ospedale Civile Cosenza, Cosenza
  - Ospedale San Giuseppe, Milan
  - Ospedale Luigi Sacco, Milan
  - Ospedale San Paolo, Milan
  - Federico II University Medical School, Naples
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Ospedale Vincenzo Monaldi, Naples
  - Seconda Universita di Napoli, Naples
  - Ospedale Civile P.F. Calvi, Noale
  - Azienda Ospedaliera Policlinico Paolo Giaccone, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Ospedale San Carlo, Potenza
  - Ospedale da Procida, Salerno

REFERENCES:
- [Background] Di Maio M, Perrone F, Chiodini P, Gallo C, Camps C, Schuette W, Quoix E, Tsai CM, Gridelli C. Individual patient data meta-analysis of docetaxel administered once every 3 weeks compared with once every week second-line treatment of advanced non-small-cell lung cancer. J Clin Oncol. 2007 Apr 10;25(11):1377-82. doi: 10.1200/JCO.2006.09.8251. PMID 17416857
- [Result] Gridelli C, Gallo C, Di Maio M, Barletta E, Illiano A, Maione P, Salvagni S, Piantedosi FV, Palazzolo G, Caffo O, Ceribelli A, Falcone A, Mazzanti P, Brancaccio L, Capuano MA, Isa L, Barbera S, Perrone F. A randomised clinical trial of two docetaxel regimens (weekly vs 3 week) in the second-line treatment of non-small-cell lung cancer. The DISTAL 01 study. Br J Cancer. 2004 Dec 13;91(12):1996-2004. doi: 10.1038/sj.bjc.6602241. PMID 15558071